CLINICAL TRIAL: NCT01587053
Title: Anti Vitamin K Therapeutic Education With INR Self Measure Device Within Children From 0 to 18 Years
Brief Title: Anti Vitamin K Therapeutic Education
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8745
Record Dates: First submitted 2012-04-12; First posted 2012-04-27 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Cardio-vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AVK: patient with AVK treatment
  Interventions: Other: therapeutic education program

INTERVENTIONS:
Other: therapeutic education program

SUMMARY:
The purpose of this study is to measure the INR (International Normalized Ratio) time percentage in the target zone (TTR: time in therapeutic range) of children benefiting from the AVK therapeutic education program.

ELIGIBILITY:
Inclusion Criteria:

* age from 0 to 18 years
* AVK prescription
* to accept participating to AVK therapeutic education program
* informed consent form of parents or legal person

Exclusion Criteria:

* parents or legal person refusal to enter in the AVK therapeutic education

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children from 0 to 18 years having AVK prescription
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
INR (International Normalized Ratio) time percentage in the target zone (TTR: time in therapeutic range) | up to 1 year

SECONDARY OUTCOMES:
Quality of life questionnaire | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Result] Abassi H, Bajolle F, Werner O, Auer A, Marquina A, Mura T, Lavastre K, Guillaumont S, Manna F, Auquier P, Bonnet D, Amedro P. Health-related quality of life correlates with time in therapeutic range in children on anticoagulants with International Normalised Ratio self-monitoring. Arch Cardiovasc Dis. 2020 Dec;113(12):811-820. doi: 10.1016/j.acvd.2020.05.022. Epub 2020 Oct 14. PMID 33069639